CLINICAL TRIAL: NCT06893731
Title: Healthcare Utilization and Economic Burden of Cardiomyopathy in China
Status: Enrolling by invitation | Type: Observational
Sponsor: China National Center for Cardiovascular Diseases (Other Government)
Responsible Party: Principal Investigator, Lei.Song,MD.&ph.D, Principal Investigator, Clinical Professor, China National Center for Cardiovascular Diseases
Other Study IDs: 2023-ZX005
Record Dates: First submitted 2024-09-27; First posted 2025-03-25 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2024-09

CONDITIONS: Cardiomyopathies; Economic Burden
MeSH Terms: conditions — Cardiomyopathies; Financial Stress

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Cardiomyopathy is the most common inherited cardiovascular disease, showing family aggregation, and it has a huge psychological and economic burden on family members. In this study, the investigators collected clinical information and costs of patients hospitalized with cardiomyopathy and establish a database to evaluate the economic burden of cardiomyopathy.

DETAILED DESCRIPTION:
This study conducted a retrospective survey of hospitalized patients with cardiomyopathy aged ≥18 years in 13 centers in China from March 1, 2017 to March1, 2022. The investigators collected demographic and clinical information as well as healthcare utilization data of patients hospitalized with cardiomyopathy so as to evaluate the economic burden of cardiomyopathy in China.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized patients with primary discharge diagnosis meeting one of the following subtypes of cardiomyopathy were enrolled, including HCM, DCM, ACM, RCM, left ventricular non-compaction, cardiac amyloidosis, Fabry disease, Pompe disease, Danon disease, and PRKAG2 cardiac syndrome.

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients hospitalized with cardiomyopathy as the primary discharge diagnosis are recruited retrospectively from multiple centers in China between March 1, 2017 and March 1, 2022.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2017-03-01 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
total cost per hospital admission | through hospitalization completion, an average of 10 days
  Total cost per hospital admissionin is total expenditures made towards a given hospital admission, including the portion paid by the health plan and any out-of-pocket costs paid by enrollees under the plan's cost sharing.The composition of the total cost of hospitalization by categorizing itemized costs into the following groups: total medical consumables cost, total diagnosis-related cost, total treatment cost (e.g., cost of operation), total Western medicine cost, total services cost, total blood and blood products cost, total traditional Chinese medicine cost, total traditional Chinese treatment cost, total rehabilitation cost, and other costs.

CONTACTS AND LOCATIONS:
Locations (1):
- Fuwai hospital, Beijing, Beijing 100037, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided